CLINICAL TRIAL: NCT00373789
Title: Refractory Urge Incontinence and Botox Injections
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: higher than anticipated rate of increased post-void residual in subjects who received botulinum toxin A injection
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Susan Meikle, MD, NICHD
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PFDN 12
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-10

CONDITIONS: Urinary Incontinence; Detrusor Overactivity; Urinary Urgency; Urge Urinary Incontinence
Keywords: Botulinum Toxin A; Urinary Incontinence; Detrusor Overactivity
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botox A (Experimental): up to two injections of 200 Units of intra-detrusor Botulinum Toxin A , which must be separated by at least eight weeks and no more than 52 weeks
  Interventions: Drug: Botulinum Toxin A, bladder detrusor muscle injection
- Placebo (Placebo Comparator): up to two injections of inactive injection (carrier saline), which must be separated by at least eight weeks and no more than 52 weeks
  Interventions: Drug: Vehicle saline as placebo

INTERVENTIONS:
Drug: Botulinum Toxin A, bladder detrusor muscle injection — 200 U provided as a total of 6 cc of the masked substance into approximately 15 to 20 different detrusor muscle sites under direct visualization. Injections will be spread out to equally cover the entire dome of the bladder, but spare the bladder trigone and ureteral orifices.
  Other Names: Botox
  Arms: Botox A
Drug: Vehicle saline as placebo — A total of 6 cc of the masked substance into approximately 15 to 20 different detrusor muscle sites under direct visualization. Injections will be spread out to equally cover the entire dome of the bladder, but spare the bladder trigone and ureteral orifices
  Arms: Placebo

SUMMARY:
The purpose of this study is to see whether Botox A (injected into the bladder muscle) can improve symptoms of urge incontinence that has not improved with usual medical treatments.

DETAILED DESCRIPTION:
Women who suffer with urge incontinence may not get relief with usual medical treatment (such as medications or behavioral techniques). We plan to enroll women with refractory urge incontinence in centers across the US. Study participants will undergo cystoscopy (telescope look into the bladder) and injection of either Botox A or placebo. If symptoms are not adequately relieved, subjects participants will receive a second injection that is Botox A. Participants are interviewed monthly by study personnel to determine symptoms and health status.

ELIGIBILITY:
Inclusion Criteria:

* Adult women
* Detrusor overactivity incontinence confirmed by urodynamic testing
* Symptoms refractory to standard first- and second-line treatments
* 6 or more urge incontinence episodes on 3-day bladder diary
* Normal neurological examination

Exclusion Criteria:

* Urinary retention
* Allergy to Botox (Botulinum Toxin A)
* Previous bladder treatment with Botox (Botulinum Toxin A) in the past year
* Pregnancy or planning pregnancy within next year
* Neurologic disease with impaired neurotransmission

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Time to recurrence of detrusor overactivity incontinence symptoms | 6 months
  To allow sufficient time for the onset of action of botulinum toxin A, the earliest outcome measurement was 60 days after injection. Failure was defined as a patient global impression of improvement (PGI-I) score of 4 or greater, the commencement of any new treatment at any time after the first injection or increased intensity of previously established treatment for DOI.

SECONDARY OUTCOMES:
Change in incontinence episode frequency by bladder diary | At 12 mos after first injection., but no less than 1 mo after second injection
  based on the 3-day bladder diary completed pre-intervention and at 4 weeks post injection. A successful within-subject outcome will be defined as >75% reduction in the frequency of urge incontinence episodes compared to the baseline frequency.
Incontinence-related and health-related quality of life | At 12 mos after first injection, but no less than 1 mo after second injection.
  measured by the Urinary Distress Inventory subscale of the PFDI/PFIQ, the PISQ, and SF-36 administered at 4 weeks after the initial injection and either prior to any re-treatment or at the completion of study participation, whichever is earlier.
Voiding dysfunction requiring catheterization | throughout 12-month study

CONTACTS AND LOCATIONS:
Overall Officials: Linda Brubaker, MD, Study Chair — Loyola University
Locations (8):
- United States (8):
  - University of Alabama, Birmingham, Alabama
  - USCD Medical Center, La Jolla, California
  - Kaiser Permanente, San Diego, California
  - Loyola University, Maywood, Illinois
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UT Southwestern, Dallas, Texas
  - Univeristy of Utah, Salt Lake City, Utah

REFERENCES:
- [Result] Brubaker L, Richter HE, Visco A, Mahajan S, Nygaard I, Braun TM, Barber MD, Menefee S, Schaffer J, Weber AM, Wei J; Pelvic Floor Disorders Network. Refractory idiopathic urge urinary incontinence and botulinum A injection. J Urol. 2008 Jul;180(1):217-22. doi: 10.1016/j.juro.2008.03.028. Epub 2008 May 21. PMID 18499184
- See also: Website of the National Institute of Child Health and Human Development, which funds the Pelvic Floor Disorders Network — http://www.nichd.nih.gov